CLINICAL TRIAL: NCT00980733
Title: Efficacy of Consumption of Micronutrient Fortified Yoghurt on Biochemical Markers, Cognitive Development, Morbidity and Physical Growth Among 6-9 Years School Going Children in Bangladesh - A Double Masked, Randomized Trial With a Concurrent Matched Control
Brief Title: Efficacy of Micronutrient Fortified Yoghurt in School Children for Health Benefits
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Annamalai University (Other)
Collaborators: Johns Hopkins Bloomberg School of Public Health (Other); Department of Community Medicine SZMC, Bogra Bangladesh (Unknown); Global Alliance for Improved Nutrition (Other)
Responsible Party: Sunil Sazawal, CMR Annamalai University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Global Alliance G#102512
Record Dates: First submitted 2009-09-18; First posted 2009-09-21 (Estimated); Last update posted 2009-09-21 (Estimated); Status verified 2009-09

CONDITIONS: Child Development; Cognitive Development; Morbidity; Physical Growth
Keywords: Micronutrients; zinc; iron; iodine; fortification; school children
MeSH Terms: interventions — Yogurt

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Fortified Yoghurt (Active Comparator): Yoghurt with fortification of Micronutrients, yoghurt fortified with 1/3rd RDA of iron, zinc, vitamin A and iodine. The salts used for fortification will be iron- Ferric pyrophosphate micronized, zinc - zinc gluconate, Iodine - Potassium Iodide, Vitamin A - Vitamin A acetate.
  Interventions: Dietary Supplement: Fortified Yoghurt
- Yoghurt (Placebo Comparator): Plain Yoghurt same as in fortified arm but without fortification
  Interventions: Dietary Supplement: Yoghurt
- Control (No Intervention): Non blinded group given no intervention

INTERVENTIONS:
Dietary Supplement: Fortified Yoghurt — The study group would receive yoghurt fortified with 1/3rd RDA of iron, zinc, vitamin A and iodine. The salts used for fortification will be iron- Ferric pyrophosphate micronized, zinc - zinc gluconate, Iodine - Potassium Iodide, Vitamin A - Vitamin A acetate.
  Arms: Fortified Yoghurt
Dietary Supplement: Yoghurt — Plain yoghurt same as in intervention group without fortification
  Arms: Yoghurt

SUMMARY:
To evaluate the efficacy of consumption of yoghurt fortified with 30% recommended dietary allowance (RDA) of essential micronutrients (iron, zinc, vitamin A and iodine) for a period of one year in comparison to same yoghurt without fortification for change in mean levels and proportion deficient for markers of status of Iron (Hemoglobin, Serum ferritin, Serum transferrin, ZnPP), Vitamin A (Plasma retinol levels), Iodine (Urinary iodine levels), Zinc (Plasma zinc), and copper (Plasma copper levels, sub sample of children); improvement in cognitive development, reduction in episodes/days of illnesses (diarrhea, pneumonia, febrile illness), hospitalizations and morbidity causing absenteeism from school and improvement in growth. Additionally to evaluate the efficacy of consumption of fortified and non fortified yoghurt (plain yoghurt) for a period of 12 months in comparison to pure control that do not receive any intervention in the improvement in cognitive development and physical growth. The main objective is to evaluate the impact of addition of micronutrients to Yoghurt and can be best addressed by RCT. The effect of taking yoghurt per se cannot be blinded so for that the investigators have included a concurrent control.

Hypothesis: Consumption of fortified yoghurt with 30% RDA of essential micronutrients (iron, zinc, vitamin A and iodine) for a period of one year will improve the micronutrient status indicators, cognitive development, and growth and reduce morbidity of children.

DETAILED DESCRIPTION:
Study population: Children aged 6-9 years both boys and girls from 6 primary schools of Gabtali town of Bogra district in Bangladesh.

Sample Size: 1200 children (400 in each group) Enrollment of eligible children and Base line information: Details of all eligible children will be obtained from the schools to be a part of the study and their parents will be contacted for an appointment either by telephone or sending a note. Consent for participation will be sought after evaluating inclusion and exclusion criteria and will be randomized to receive either fortified or non fortified yoghurt, similarly consent will be obtained from the parents of children from the non yoghurt area who will not be given any intervention. Baseline information on socioeconomic information, retrospective morbidity information of the child for the last 15 days, hospitalization, hygiene and sanitation information will be recorded. Baseline clinical assessments and anthropometric measurements will be conducted. 5 ml of venous blood sample (approx. one spoonful of blood) and mid stream urine sample will be obtained by a trained nurse/technician employed by the project. Developmental assessments measuring children's intelligence and executive functioning (WISC, KCPT, WCST) will be conducted using standardized tests. Blood/urine sampling will not be done for the children in the pure control group (no intervention).

Randomization and blinding: Randomization schedule will be drawn using randomization by permuted blocks of fixed length which is appropriate for double blind studies.

Intervention and Follow-up: For the yoghurt group, the intervention would be supplied in a disposable 80 g cup. Computer labels will be generated on a daily basis with identification information and the allocated code printed on it for all the enrolled children in the database and the appropriate yoghurt cups will be labeled for each child. The labeled yoghurt cups will be then handed over to the school supervisor to deliver to the student in his/her supervision during lunch break of the school. Children will receive the intervention for a period of 12 months. Children from the matched control in the non-yoghurt area will not receive any intervention.

Mid Study data collection: Similar to the baseline, anthropometric measurements will be done and again a 5ml blood sample (approx one spoonful of blood) will be obtained to assess the difference in the markers at baseline and mid study. Blood/urine sampling will not be done for children in the pure control.

End Study data collection: An end study similar to the baseline, anthropometric measurements will be taken and again a 5ml blood sample (approx one spoonful of blood) will be obtained to assess the difference in the markers at baseline and end study. Blood/urine sampling will not be done for the children in the pure control (no intervention group). Detailed developmental assessments using a battery of computerized neuropsychological (CANTAB) and cognition tests (WISC, K-CPT and WCST) will be conducted. Academic achievement will be assessed using school report cards.

Intervention Groups: There will be one study group with one control group. Both the groups would receive yoghurt in a 80 g cup. The study group would receive yoghurt fortified with 1/3rd RDA of iron, zinc, vitamin A and iodine.

ELIGIBILITY:
Inclusion Criteria:

* children aged between 6 to 9 yrs of age,
* enrolled in the school,
* not severely malnourished requiring rehabilitation and micronutrient supplement, AND
* consent to participate.

Inclusion is only based on age and locale: 6-9 years in Gabtali schools and both genders will be enrolled.

Exclusion Criteria:

* children who are severely malnourished and requiring hospitalization.

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1325 (Estimated)
Dates: Start 2008-09; Primary Completion 2010-04 (Estimated); Study Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
Morbidity | 0 months, 6 months, 12 months
Growth | 0 months, 6 months, 12 months
Development | 0 months, 6 months, 12 months
School performance | 0 months, 6 months, 12 months
Status Indicators for iron, zinc, vitamin A and iodine | 0 months, 6 months, 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Community Medicine, SZMC, Bogra, Bangladesh

REFERENCES:
- [Background] Winichagoon P, McKenzie JE, Chavasit V, Pongcharoen T, Gowachirapant S, Boonpraderm A, Manger MS, Bailey KB, Wasantwisut E, Gibson RS. A multimicronutrient-fortified seasoning powder enhances the hemoglobin, zinc, and iodine status of primary school children in North East Thailand: a randomized controlled trial of efficacy. J Nutr. 2006 Jun;136(6):1617-23. doi: 10.1093/jn/136.6.1617. PMID 16702330
- [Background] Grantham-McGregor SM, Ani CC. The role of micronutrients in psychomotor and cognitive development. Br Med Bull. 1999;55(3):511-27. doi: 10.1258/0007142991902583. PMID 10746342
- [Derived] Sazawal S, Habib A, Dhingra U, Dutta A, Dhingra P, Sarkar A, Deb S, Alam J, Husna A, Black RE. Impact of micronutrient fortification of yoghurt on micronutrient status markers and growth - a randomized double blind controlled trial among school children in Bangladesh. BMC Public Health. 2013 May 28;13:514. doi: 10.1186/1471-2458-13-514. PMID 23714325